CLINICAL TRIAL: NCT05145140
Title: A Clinical Intervention Study of Tangningtongluo on Diabetic Foot Ulcer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNTL on diabetic foot ulcer
Record Dates: First submitted 2021-09-02; First posted 2021-12-06 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — tangningtongluo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standardized Western Medicine Treatment Group (Active Comparator): All participants undergo a similar treatment protocol for the diabetic foot, based on the Infectious Diseases Society of America (IDSA).
  Interventions: Drug: Standardized Western Medicine Treatment
- Standardized Western Medicine Treatment +TNTL tablet+TNTL cream Group (Experimental): Treatment with TNTL tablets:the oral administration of TNTL tablets, 4 tablets each time, 3 times a day. Treatment with TNTL cream: topical application of sterile TNTL cream on the wound surface, the dressing is continuously changed according to the wound healing.
  Interventions: Drug: Standardized Western Medicine Treatment; Drug: Tangningtongluo tablet and cream
- Standardized Western Medicine Treatment +TNTL tablet Group (Experimental): Treatment with TNTL tablets:the oral administration of TNTL tablets, 4 tablets each time, 3 times a day.
  Interventions: Drug: Standardized Western Medicine Treatment; Drug: Tangningtongluo tablet
- Standardized Western Medicine Treatment +TNTL cream Group (Experimental): Treatment with TNTL cream: topical application of sterile TNTL cream on the wound surface, the dressing is continuously changed according to the wound healing.
  Interventions: Drug: Standardized Western Medicine Treatment; Drug: Tangningtongluo cream

INTERVENTIONS:
Drug: Standardized Western Medicine Treatment — Standardized Western Medicine Treatment includes hypoglycemic, debridement and anti infection treatments.
  Other Names: Classic Diabetic Foot Ulcer treatment
Drug: Tangningtongluo tablet and cream — Tangningtongluo(TNTL) , a traditional botanical ethnic medicine, composed of plantain, honeysuckle, agrimony, etc. It is famous for its effects of promoting blood circulation, dredging collaterals, reducing thirst and lowering glucose.There are two dosage forms: tablet and cream.
  Other Names: Tangningtongluo Pian and Tangningtongluo Gao
  Arms: Standardized Western Medicine Treatment +TNTL tablet+TNTL cream Group
Drug: Tangningtongluo tablet — Tangningtongluo(TNTL) , a traditional botanical ethnic medicine, composed of plantain, honeysuckle, agrimony, etc. It is famous for its effects of promoting blood circulation, dredging collaterals, reducing thirst and lowering glucose.The participants in this arm use tablet.
  Other Names: Tangningtongluo Pian
  Arms: Standardized Western Medicine Treatment +TNTL tablet Group
Drug: Tangningtongluo cream — Tangningtongluo(TNTL) , a traditional botanical ethnic medicine, composed of plantain, honeysuckle, agrimony, etc. It is famous for its effects of promoting blood circulation, dredging collaterals, reducing thirst and lowering glucose.The participants in this arm use cream.
  Other Names: Tangningtongluo Gao
  Arms: Standardized Western Medicine Treatment +TNTL cream Group

SUMMARY:
Purpose and significance:With the increasing incidence of Diabetes mellitus (DM), the incidence rate of Diabetic Foot (DF) is raised. DF is a foot infection, ulceration and / or deep tissue destruction caused by nerve abnormalities and varying degrees of vascular lesions in DM patients. The high incidence, disability and mortality rate of DF make it urgent to explore new ways to improve the cure rate, reduce the burden and elevate the quality of life. Previous studies have confirmed that traditional Miao ethic medicine Tangningtongluo(TNTL) can improve the remission rate of diabetes mellitus and diabetic foot disease, but the clinical research evidence is not sufficient. This study aims to provide effective clinical evidence for the treatment of diabetic foot patients with TNTL by observing growth rate of wound, prognosis and outcome.

Methods: From September 2021 to March 2023, a total of 80 diabetic foot ulcer patients admitted to Department of Endocrinology and Metabolism at the Affiliated Hospital of Nantong University were recruited. Participants are randomized in a ratio of 1: 1: 1:1 into four treatment groups of 20 participants: (i) standardized western medicine treatment group, (ii) standardized western medicine treatment+TNTL tablet+TNTL cream group , (iii) standardized western medicine treatment+TNTL tablet group, and (iiii) standardized western medicine treatment+TNTL cream group. Treatment with TNTL tablets: the oral administration of TNTL tablets, 4 tablets each time, 3 times a day. Treatment with TNTL cream: topical application of sterile TNTL cream on the wound surface, the dressing is continuously changed according to the wound healing. Anthropometric parameters, serum biochemical index, glycosylated hemoglobin, urinary microalbumin/creatinine ratio, islet-specific autoantibodies(ISAs), fat mass, and islet β-cell function were measured. The healing stage of the wound surface and the growth degree of granulation tissue were graded, and the time required for wound repairing to each healing stage was observed.

Type of study: randomized controlled, prospective,intervention study.

DETAILED DESCRIPTION:
From September 2021 to March 2023, a total of 80 diabetic foot ulcer patients admitted to Department of Endocrinology and Metabolism at the Affiliated Hospital of Nantong University were recruited. Participants are randomized in a ratio of 1: 1: 1:1 into four treatment groups of 20 participants: (i) standardized western medicine treatment group, (ii) standardized western medicine treatment+TNTL tablet+TNTL cream group , (iii) standardized western medicine treatment+TNTL tablet group, and (iiii) standardized western medicine treatment+TNTL cream group. Treatment with TNTL tablets: the oral administration of TNTL tablets, 4 tablets each time, 3 times a day. Treatment with TNTL cream: topical application of sterile TNTL cream on the wound surface, the dressing is continuously changed according to the wound healing. Anthropometric parameters, serum biochemical index, glycosylated hemoglobin, urinary microalbumin/creatinine ratio, islet-specific autoantibodies(ISAs), fat mass, and islet β-cell function were measured. The healing stage of the wound surface and the growth degree of granulation tissue were graded, and the time required for wound repairing to each healing stage was observed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes mellitus
* Clinical diagnosis of Diabetic Foot Ulcer

Exclusion Criteria:

* Type 1 diabetes mellitus(T1DM), special type of diabetes, gestational diabetes mellitus, drug-induced hyperglycemia
* TNTL allergy
* Chronic kidney failure（eGFR≤30ml/min/1.73cm2）, severe liver function damage (transaminase ≥ 3 times the normal value), acute or chronic pancreatitis, autoimmune disease, malignant tumors
* Recent acute complications of type 2 diabetes mellitus（ketoacidosis, hyperosmolar nonketotic diabetic coma, lactic acidosis etc.）or other emergency situations
* History of using glucocorticoids and immunosuppressants
* Mental illness and cognitive dysfunction or poor compliance, unable to take medication as required
* Malignant ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Decrease area of wound healing due to Diabetic Foot Ulcer | 12 weeks
  Assessment the decrease of whole area of diabetic foot ulcers. The unit is square centimeters .
Decrease of depth of ulcer involve the deep fascia. | 12 weeks
  Measurement of depth of ulcer involve the deep fascia. The unit is millimeters.
Amputation Rate | 12 weeks
  The difference of end-stage amputation rates between the experimental group and the control group were evaluated by the arterial and venous blood circulation of the lower limbs
Diabetic Foot Ulcer relapse rate | 12 weeks
  The relapse of Diabetic Foot Ulcers is a common complication in the advanced stage of DFU. The difference of treatment between the experimental group and the control group indicates that the prognosis is variability.

SECONDARY OUTCOMES:
Fasting glucose | 12 weeks
  10 hours after fasting peripheral blood glucose level, and the unit is mmol/L
2-H postload glucose | 12 weeks
  2 hours after peripheral blood glucose level eating 75g glucose or 100g steamed bread, and the unit is mmol/L
BMI Index | 12 weeks
  The calculation formula of Body Mass Index is: BMI = weight ÷ height 2. (weight in kilograms; height in meters.)
WHR Index | 12 weeks
  Waist to hip ratio (WHR) = waist / hip.Waist circumference or minimum waist circumference shall be used for measurement, and evaluation of WHR is an important value to central obesity.
Islet B cell function | 12 weeks
  The ability of islet B cells to secrete insulin was reflected by the level of C peptide, which is measured after fasting. The unit is ng/dL .
interleukin-6(IL-6) | 12 weeks
  Determine the level of interleukin-6(IL-6) in peripheral blood by ELISA, the unit is ng/L.
tumour necrosis factor-α(TNF-α) | 12 weeks
  Determine the level of TNF-α in peripheral blood , the unit is ng/ml.
C-reactive protein(CRP) | 12 weeks
  Determine the level of C-reactive protein(CRP) in peripheral blood , the unit is μg/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yunjuan, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No